CLINICAL TRIAL: NCT05520619
Title: Tislelizumab Plus Induction Chemotherapy Followed by Concurrent Chemoradiotherapy for Patients with Locally Advanced Esophageal Squamous Cell Carcinoma: a Phase II, Randomized Trial (EC-CRT-002)
Brief Title: Combination of Tislelizumab and Chemoradiotherapy in Esophageal Cancer (EC-CRT-002)
Acronym: EC-CRT-002
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Jieyang People's Hospital (Other)
Responsible Party: Principal Investigator, Mian XI, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2022-216-02
Record Dates: First submitted 2022-08-21; First posted 2022-08-30 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma; Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Induction chemotherapy; Definitive chemoradiotherapy; Tislelizumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — TP protocol; Paclitaxel; tislelizumab; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tislelizumab plus CRT with maintenance (Experimental): Patients will receive 2 cycles of 3-weekly schedule of induction chemotherapy, consisting of paclitaxel 135-175 mg/m2, cisplatin 75 mg/m2, and tislelizumab 200mg on day 1 prior to CRT. Then all patients will receive standard fractionation radiation therapy scheme: 50.4 Gy in 28 fractions, concurrently with paclitaxel 45mg/m2 and cisplatin 25 mg/m2 once weekly for 5 weeks and 2 cycles of tislelizumab. Patients in Arm A will receive 12 additional cycles of tislelizumab after the completion of radiotherapy.
  Interventions: Drug: Paclitaxel, Cisplatin; Drug: tislelizumab; Radiation: Radiotherapy
- Tislelizumab plus CRT without maintenance (Experimental): Patients will receive 2 cycles of 3-weekly schedule of induction chemotherapy, consisting of paclitaxel 135-175 mg/m2, cisplatin 75 mg/m2, and tislelizumab 200mg on day 1 prior to CRT. Then all patients will receive standard fractionation radiation therapy scheme: 50.4 Gy in 28 fractions, concurrently with paclitaxel 45mg/m2 and cisplatin 25 mg/m2 once weekly for 5 weeks and 2 cycles of tislelizumab. Patients in Arm B will receive 4 cycles of tislelizumab in total.
  Interventions: Drug: Paclitaxel, Cisplatin; Drug: tislelizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin — Patients received 2 cycles of induction chemotherapy with paclitaxel/cisplatin (paclitaxel 135-175mg/m2 and cisplatin 75 mg/m2) prior to radiotherapy. Then patients will receive paclitaxel 45mg/m2 and cisplatin 25 mg/m2 once weekly for 5 weeks during radiotherapy.
  Other Names: Taxol
Drug: tislelizumab — Patients received tislelizumab 200 mg every 3 weeks for 16 cycles in Arm A and 4 cycles in Arm B.
Radiation: Radiotherapy — All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is 50.4 Gy in 28 fractions over 5-6 weeks.
  Other Names: intensity-modulated radiotherapy

SUMMARY:
Definitive chemoradiotherapy (CRT) is the standard treatment option for unresectable locally advanced esophageal cancer (EC). However, as high as more than 40% of EC patients experienced locoregional recurrence after concurrent CRT. Immunotherapy targeting the PD-1/PD-L1 checkpoints has demonstrated promising activity in advanced EC. Recently, the combination of immunotherapy with CRT has emerged as a promising strategy to improve clinical outcomes in EC. The aim of this study was to evaluate whether the efficacy of tislelizumab (an anti-PD-1 antibody) plus induction chemotherapy followed by concurrent chemoradiotherapy would achieve a ≥71% 1-year progression-free survival rate, surpassing the historical 56% rate (NCT02403531) in patients with locally advanced esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
A total of 114 patients with unresectable, locally advanced ESCC will be randomized to receive either tislelizumab plus induction chemotherapy followed by concurrent CRT and then 12 additional cycles of tislelizumab (Arm A) or tislelizumab plus the same induction and concurrent regimen without the maintenance of tislelizumab (Arm B).

Patients will receive 2 cycles of 3-weekly schedule of induction chemotherapy, consisting of paclitaxel 135-175 mg/m2, cisplatin 75 mg/m2, and tislelizumab 200mg on day 1 prior to CRT. Then all patients will receive standard fractionation radiation therapy scheme: 50.4 Gy in 28 fractions, concurrently with paclitaxel 45mg/m2 and cisplatin 25 mg/m2 once weekly for 5 weeks and 2 cycles of tislelizumab. Patients in Arm A will receive 12 additional cycles of tislelizumab after the completion of CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Locally advanced, and absence of hematogenous metastasis disease, confirmed by endoscopic ultrasound (EUS) and PET-CT scan (according to UICC TNM version 8);
3. Not suitable for surgery (either for medical reasons or patient's choice);
4. Age at diagnosis 18 to 70 years;
5. No prior cancer therapy;
6. Estimated life expectancy >6 months;
7. Eastern Cooperative Oncology Group performance status ≤ 2
8. No history of concomitant or previous malignancy;
9. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥4.0×109/L, absolute neutrophil count (ANC) ≥1.5×109/L; b. platelets ≥100×109/L; c. hemoglobin ≥9g/dL; d. serum albumin ≥2.8g/dL; e. total bilirubin ≤1.5×ULN, ALT, AST and/or AKP ≤2.5×ULN; f. serum creatinine ≤1.5×ULN or creatinine clearance rate >60 mL/min;
10. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Patients with hematogenous metastasis disease at diagnosis;
3. Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of Toripalimab, and the chemotherapeutic drugs paclitaxel or cisplatin;
4. Patients who have a preexisting or coexisting bleeding disorder;
5. Female patients who are pregnant or lactating;
6. Inability to provide informed consent due to psychological, familial, social and other factors;
7. Presence of CTC grade ≥ 3 peripheral neuropathy;
8. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer
9. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
10. Patients who cannot tolerate chemoradiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia.
11. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
12. A history of interstitial lung disease or non-infectious pneumonia;
13. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  Two-year follow-up from the date of randomization to the date of disease progression or last follow-up

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 24 months.
  Two-year follow-up from the enrollment to the date of death from any cause or date of lost follow-up
Duration of response | From date of first CR/PR to the date of first PD according to RECIST criteria, assessed up to 24 months
  From the date of first CR/PR to the date of first PD.
Clinical complete response | Three months after the treatment (plus or minus 7 days)
  RECIST (Response Evaluation Criteria in Solid Tumors) criteria was used to determine the tumor response. Tumor response was evaluated 3 months after the completion of treatment based on CT or PET-CT scans, and endoscopy with biopsies.
Treatment-related adverse events | From date of randomization until the date of last follow-up, assessed up to 12 months.
  Incidence of treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
PD-L1 expression | From date of randomization until the date of last follow-up, assessed up to 24 months.
  To investigate the impact of PD-L1 expression on clinical response and survival.
ctDNA at baseline, during, and after treatment | From date of randomization until the date of last follow-up, assessed up to 24 months.
  To investigate the impact of dynamic change of ctDNA on clinical response and survival.
CD8 expression at baseline | From date of randomization until the date of last follow-up, assessed up to 24 months.
  To investigate the impact of CD8 expression on clinical response and survival.
Tumor mutational burden at baseline | From date of randomization until the date of last follow-up, assessed up to 24 months.
  To investigate the impact of tumor mutational burden by whole-exome sequencing on clinical response and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Mian Xi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Background] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801